CLINICAL TRIAL: NCT01392950
Title: Clinical Performance of the Clariti Monthly Contact Lens for Daily Wear
Brief Title: Clinical Study of Clariti Monthly Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sauflon Pharmaceuticals Ltd (Industry)
Responsible Party: Howard Griffiths, Sauflon Pharmaceuticals Limited
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: S10-491
Record Dates: First submitted 2011-07-06; First posted 2011-07-13 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Hyperopia; Myopia
Keywords: silicone hydrogel contact lenses for daily wear
MeSH Terms: conditions — Hyperopia; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Optix Aqua (Active Comparator): Compare safety and efficacy using OptiFree Replenish solution
  Interventions: Device: Air Optix Aqua
- Clariti (Active Comparator): Compare safety and efficacy of the lens using OptiFree Replenish solution
  Interventions: Device: Clariti

INTERVENTIONS:
Device: Air Optix Aqua — Lenses will be worn on a daily wear basis (ie. removed at night and stored in solution) and worn in the normal way. Lenses will be replaced each month. Lenses should be worn for a minimum of six hours a day, four days a week. The lenses are also to be worn for a minimum of two hours before attending all follow-up visits.
  Arms: Air Optix Aqua
Device: Clariti — Lenses will be worn on a daily wear basis (ie. removed at night and stored in solution) and worn in the normal way. Lenses will be replaced each month. Lenses should be worn for a minimum of six hours a day, four days a week. The lenses are also to be worn for a minimum of two hours before attending all follow-up visits.
  Arms: Clariti

SUMMARY:
A clinical study report follows; this clinical study evaluated the safety and efficacy of SAUFLON CLARITI Soft Silicone Hydrogel Contact Lens with UV Blocker by comparison with Air Optix Aqua silicone hydrogel contact lenses (Ciba Vision Inc.).

Subjects used OptiFree Replenish solution (Alcon Laboratories Inc.) for daily lens maintenance, care and storage.

DETAILED DESCRIPTION:
1.1 Study characteristics This study evaluated the safety and efficacy of Clariti Monthly silicone hydrogel contact lenses (Sauflon Pharmaceuticals Limited) by comparison with Air Optix Aqua silicone hydrogel contact lenses (Ciba Vision Inc.). Subjects used OptiFree Replenish solution(Alcon Laboratories Inc.) for daily lens maintenance, care and storage.

The key study features were as follows:

1. Three months duration.
2. Seven investigator sites.
3. Daily wear soft (hydrophilic) silicone hydrogel contact lenses, replaced on a monthly basis: Clariti Monthly and Air Optix Aqua. OptiFree Replenish was used as a care system by all subjects.
4. A total of 95 subjects were enrolled, and 94 subjects accounting for 188 eyes were dispensed lenses. This group was randomized into 64 test subjects (128 eyes)and 30 control subjects (60 eyes).
5. Of the 64 test subjects, 56 (87.5%) completed three months of use. Of the 30 control subjects, 29 (96.7%) completed three months of use.
6. No eyes remained active at the end of the study.
7. There were no adverse reactions.

1.2 Study period The study was conducted over three months of wear. Subjects were examined initially,and at five follow-up visits after one week, two weeks, four weeks, eight weeks and 12 weeks. Study visits commenced on September 6, 2010 and were completed on March 16, 2011.

1.3 Demographics Seven investigator sites dispensed 64 test subjects (128 eyes) who used Clariti Monthly as their contact lens during the work. Also enrolled were 30 control subjects (60 eyes)who used Air Optix Aqua as their contact lens during the work. All recruited subjects were existing contact lenses wearers.

Of the 64 test subjects, 56 (87.5%) completed three months of use and eight (12.5%)were discontinued. Of the 30 control subjects, 29 (96.7%) completed three months of use and one (3.4%) was discontinued.

The enrolled control group was made up of 22 females (73%) and eight males (27%) with an age range from 19 to 63 years (mean 35.6 years). The enrolled test group was composed of 41 females (63%) and 24 males (37%) with an age range from 17 to 62 years (mean 32.8 years). One ineligible subject (age 17 years) was enrolled and assigned to the test group but was not dispensed lenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will only be eligible for the study if:

  1. They are 18 years of age and above.
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They agree not to participate in other clinical research for the duration of this study.
  5. They can attain at least 6/9 in each eye with the study contact lenses.
  6. They have successfully worn contact lenses within six months of starting the study.
  7. They can be fitted with spherical soft contact lenses within the power range available.

Exclusion Criteria:

* Subjects will not be eligible if:

  1. They have an ocular disorder which would normally contra-indicate contact lens wear.
  2. They have a systemic disorder which would normally contra-indicate contact lens wear.
  3. They are using any topical medication such as eye drops or ointment.
  4. They have glaucoma (high pressure in the eye), have had cataract surgery or a history of recurring abrasions.
  5. They have had corneal refractive surgery.
  6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
  7. They are pregnant or lactating.
  8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
  9. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 19 Years to 63 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Overall subjective acceptance | 3 months
  The results of this study showed the safety, acceptability and substantial equivalence of the Sauflon CLARITI (somofilcon A) Soft Silicone Hydrogel Contact Lens with UV Blocker to the predicate device for its intended use.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD, Principal Investigator — MCOptom FAAO FBCLA
Locations (1):
- Eurolens Research Faculty of Life Sciences The University of Manchester, Manchester, Manchester, United Kingdom